CLINICAL TRIAL: NCT03406910
Title: Egg Intake and Risk of Type 2 Diabetes in a Low Meat Intake Population
Brief Title: Egg Intake and Risk of Type 2 Diabetes
Acronym: ES
Status: Completed | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Professor of Nutrition and Epidemiology, Loma Linda University
Other Study IDs: 2140392
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Type 2 Diabetes; Heart Diseases
Keywords: egg; meat; western diet; type 2 diabetes; Adventist Health Study; Vegetarian cohort; Adventist
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Seventh day Adventist adults: Seventh day Adventist adults recruited from the USA and Canada. Approximately 65% female and 35% male. Composed of participants with different dietary patterns and a wide variation in egg and meat intake ranging from non-consumptive to daily consumption.

SUMMARY:
This is a longitudinal study that will collect demographic, anthropometric and dietary data to determine the relationships between meat and egg intake and the incidence of Type 2 Diabetes.

DETAILED DESCRIPTION:
Subjects of the Adventist Health Study who are non-diabetic will provide demographic, anthropometric and dietary data at baseline. Meat and egg intake will be assessed with a validated quantitative food frequency intake questionnaire. The relationship between meat and egg intake and the incidence of Type 2 Diabetes will be determined using multivariate-adjusted logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* AHS 2 Participants who filled out Hospital History Questionnaire version 3 or 5 Age > 30 years

Exclusion Criteria:

* Subjects with missing values in dietary variables were excluded from the analytic sample,
* missing gender
* age < 30 years
* improbable questionnaire response patterns
* extremes of BMI (less than 16 or greater than 60)
* estimated energy intake (less than 500 or greater than 4,500 kcal/d)
* existing cases of type 1 or type 2 diabetes at baseline
* inconsistent reports of T2D between HHQ version 3 and 5

Min Age: 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The AHS-2 is a prospective cohort of >96,000 Seventh-day Adventist adults recruited from the USA and Canada between February 2002 and May 2007. Designed primarily to examine associations between diet and health outcomes, the study is composed of approximately 65% females and 27% blacks. Recruitment and data collection methods for the parent cohort have been described previously. The cohort is composed of participants with different dietary patterns and a wide variation in egg and meat intake ranging from non-consumption to daily consumption. Approval for the AHS-2 study was obtained from the Loma Linda University Human Subjects Committee Institutional Review Board and written informed consent was acquired from all AHS-2 participants upon enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 55851 (Actual)
Dates: Start 2015-02-13 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Risk for Type 2 Diabetes (T2D) in subjects who consume different frequencies/amounts of eggs and meat. | Change between baseline and 5 Years of follow up
  Validated quantitative food frequency questionnaire that compares risk of T2D in subjects who consume different frequencies /amounts of egg and meat and physician diagnosis of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No